CLINICAL TRIAL: NCT06438926
Title: Prevalence of Dental Caries in Patients With Dental Crowding
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Reem Mohamed Mossaad, Principal investigator, Cairo University
Other Study IDs: Caries with dental crowding
Record Dates: First submitted 2024-05-20; First posted 2024-06-03 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Caries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Dental crowding causes limited access for the toothbrush, and the natural cleansing effect of the teeth by the tongue and saliva is also limited. This malposition allows for prolonged food accumulation, bacterial and plaque retention, which are important factors for the initiation and progression of dental caries.

DETAILED DESCRIPTION:
Dental crowding causes limited access for the toothbrush, and the natural cleansing effect of the teeth by the tongue and saliva is also limited. This malposition allows for prolonged food accumulation, bacterial and plaque retention, which are important factors for the initiation and progression of dental caries .

According to the World Health Organization, the main dental problems should be subjected to periodic epidemiological surveys. Knowledge of a population's epidemiological situation is vital for planning and providing prevention and treatment services .

However, only few studies investigated the correlation between caries and crowding.Yet, their findings were inconsistent and still contradictory.

Previous systematic review concluded that there is no reliable evidence regarding the association between dental caries and crowding and further studies with adequate sample size are required. Another systematic review found an association between caries and crowding but only in the adolescent group .

As caries is a preventable disease, improving the understanding of this possible association would be beneficial for dental practitioners, public health policy makers and the general population as it will help in the application of medical model.

This Cross-sectional study can detect one of predictors of dental caries early as crowding so the dentists can prohibit future carious lesions & help in caries prevention through orthodontic treatment & proper oral hygiene measures.

ELIGIBILITY:
Inclusion Criteria:

* Young adults range from 12-30 years.
* Females or Males.
* Anterior dental crowding.

Exclusion Criteria:

* Patients undergoing orthodontic treatment.
* Patients who have any missing anterior teeth.
* Patients who have any physical or mental disabilities.

Ages: 12 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Young adults range from 12-30 years,Females or Males with anterior dental crowding.
Sampling Method: Probability Sample
Enrollment: 325 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Dental Caries | throughout study completion an average of 1 year
  DMF index developed by WHO health organization using numbered scores

REFERENCES:
- [Background] Hafez HS, Shaarawy SM, Al-Sakiti AA, Mostafa YA. Dental crowding as a caries risk factor: a systematic review. Am J Orthod Dentofacial Orthop. 2012 Oct;142(4):443-50. doi: 10.1016/j.ajodo.2012.04.018. PMID 22999666
- [Background] Caplin JL, Evans CA, Begole EA. The Relationship between Caries and Malocclusion in Chinese Migrant Workers' Children in Shanghai. Chin J Dent Res. 2015;18(2):103-10. PMID 26167548